CLINICAL TRIAL: NCT05578157
Title: MENDiP: Measurements of Overnight Penile Temperature to Evaluate Nocturnal Erection Detection in Patients With Absence of Erectile Functioning After Robot-assisted Radical Prostatectomy
Acronym: MENDiP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Hille Torenvlied, MSc., St. Antonius Hospital
Other Study IDs: ABR: 82813
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Erectile Dysfunction; Erectile Dysfunction Following Radical Prostatectomy
Keywords: Erectile Dysfunction; Nocturnal erection; RigiScan; Penile temperature
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Age 55 - 60 years
  Interventions: Diagnostic Test: Feeling Hot sensor
- Group 2: Age 60 - 65 years
  Interventions: Diagnostic Test: Feeling Hot sensor
- Group 3: Age 65 - 70 years
  Interventions: Diagnostic Test: Feeling Hot sensor

INTERVENTIONS:
Diagnostic Test: Feeling Hot sensor — The Feeling Hot sensor is a proof-of-concept system, which can measure overnight penile, thigh and air temperature.

SUMMARY:
Nocturnal erection detection with the outdated RigiScan is the golden standard for erectile dysfunction (ED) nature differentiation. The Staying Hot and Feeling Hot study have shown that nocturnal erection detection is feasible with patient-friendly overnight penile temperature measurements. The question has arisen whether the penile temperature methodology is also capable to detect the absence of nocturnal erections, which is essential for clinical implementation in erectile dysfunction diagnostics. The objective of the MENDiP-study is to determine the feasibility to detect the absence of nocturnal erections with overnight penile temperature sensors. Furthermore, the MENDiP study functions as a first pilot trial to investigate the effect of age on the penile temperature during nocturnal erections in test subjects with normal erectile functioning. This is done in an observational study with a longitudinal design in which pre- and postoperative ambulatory overnight measurements are performed in patients, aged 55 - 70 years with preoperative normal sexual functioning, undergoing a non- or unilateral nerve-sparing robot assisted radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative measurement:

   * Aged 55 - 70 years
   * Prostatecancer patients undergoing a non-/unilateral-nerve-sparing radical prostatectomy (RARP)
   * Pre-operative IIEF-5 score > 21
2. Postoperative measurement

   * Inclusion criteria of pre-operative measurement
   * Preoperative penile temperature increase during first nocturnal erection of minimally 0.4 degrees Celsius
   * Post-operative IIEF-5 score < 12 with absence of morning erections

Exclusion Criteria:

* Test subjects who are unwilling to sign informed consent
* Test subjects with erectile dysfunction before RARP (IIEF-5 score of below 22)
* (History of) sickle cell aneamia, atherosclerosis and diabetes type I or II. These conditions might influence penile blood circulation and therefore the accuracy of the study outcomes.
* (History of) REM-sleep behavior disorder or other sleep disorders such as restless legs syndrome, insomnia, and sleep apnea
* Usage of sleeping pills or benzodiazepines.
* Postoperative results will be excluded from the study in case of presence of nocturnal erections according to the RigiScan data.

Ages: 55 Years to 70 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Fifteen patients, aged 55 - 70 years, who will undergo a non- or unilateral-nerve-sparing robot assisted radical prostatectomy will be included in case preoperative normal erectile functioning and postoperative complete impotence at three months after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-01-18 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-10-10 (Estimated)

PRIMARY OUTCOMES:
Detectability absence nocturnal erections | 9 hours
  Visual detectability of the presence and absence of nocturnal erections in overnight penile temperature measurements
Penile temperature REM-sleep | 9 hours
  Maximal variation in penile temperature during REM-sleep in case of presence and absence of nocturnal erections
Penile temperature nocturnal erection | 9 hours
  Maximal variation in penile temperature during nocturnal erections in men aged 55 - 70 years

OTHER OUTCOMES:
Demographic data | 1 year
  age, BMI, surgeries, comorbidities (diabetes, hypertension, hyperlipidemia), medication, status of smoking and alcohol consumption

CONTACTS AND LOCATIONS:
Overall Officials: Jack Beck, dr., MD, Principal Investigator — Urologist
Locations (1):
- St. Antonius Ziekenhuis, Nieuwegein, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No